CLINICAL TRIAL: NCT01789034
Title: Incidence and Predictors of Difficult Intubation Adopting an Institutional Algorithm Glidescope Based: a Cohort Study
Brief Title: Difficult Intubation With Glidescope Video Laryngoscope
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Principal Investigator, Massimo Lamperti, MD, Neuroanesthesia Department, Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta
Other Study IDs: Besta-2012-01
Record Dates: First submitted 2013-02-08; First posted 2013-02-11 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Difficult Intubation; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A prospective observational study on predictors available and on variables of difficult intubation adopting Gliscope video laryngoscope routinely.

Primary hypothesis of the current study is that the rate of difficult intubation with Glidescope is low and multiple predictors interact favorably in anticipating difficulties.

DETAILED DESCRIPTION:
All possible factors involved in difficult intubations were included in this prospective analysis.

Main predictors were considered: time to Cormack Lane using Glidescope intubation, Cormack Lane score, experience of the operator (staff or resident), number of bag mask ventilation, number of intubation attempts.

ELIGIBILITY:
Inclusion Criteria:

* any patient up to ASA4 eligible for intubation for neurosurgical procedures
* any anesthesiologist in charge for GA

Exclusion Criteria:

* children
* patient not suitable for clinical evaluation of predictors for difficult intubation (ie. Parkinson's disease)

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing neurosurgical procedures eligible for intubation in a tertiary neurosurgical centre
Sampling Method: Non-Probability Sample
Enrollment: 2600 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
incidence of difficult intubation using Adnet score modified | 3 years
  Difficult intubation in the current study is measured using Adnet score including the number of laryngoscopies

SECONDARY OUTCOMES:
incidence of difficult intubations in novices vs experts and complication in the overall cohort | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Cortellazzi, MD, Principal Investigator — Istituto Nazionale Neurologico Carlo Besta
Locations (1):
- Istituto Neurologico Besta, Milan, Italy